CLINICAL TRIAL: NCT06684652
Title: Efficacy and Safety Evaluation of Targeted Biopsy Plus Sextant Biopsy in Diagnosis of Prostate Cancer: a Randomized Controlled Trial
Brief Title: Evaluation of Targeted Biopsy Plus Sextant Biopsy in Diagnosis of Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, LIU Yi, Associate chief physician, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TB+6SB_01
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Randomized controlled trial; Targeted biopsy; Systematic biopsy; Sextant biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3TB+6SB group (Experimental): For each predefined mpMRI suspicious lesion, urologists firstly obtained three-core TB from the lesion within the mpMRI suspicious lesion. Then urologists obtained sextant six-core SB.
  Interventions: Procedure: 3TB+6SB
- 3TB+12SB group (Experimental): For patients in the 3TB+12SB group, urologists firstly obtained three-core TB from the lesion within the mpMRI suspicious lesion. Then urologists obtained fore-zone 12-core SB.
  Interventions: Procedure: 3TB+12SB

INTERVENTIONS:
Procedure: 3TB+6SB — The biopsy procedure was conducted by a highly skilled and experienced urologist who specializes in performing prostate biopsies. Prophylactic antibiotics were routinely used both before and one day prior to scheduled surgery. Each patient was placed in the left lateral position or lithotomy position. The ultrasound equipment used included a color Doppler ultrasound diagnostic instrument (Hitachi HiVision, Philips Epiq 7), transrectal probes, and corresponding puncture needle guns. Color Doppler examination was performed from the base to the apex. For each predefined mpMRI suspicious lesion, urologists firstly obtained three-core TB from the lesion within the mpMRI suspicious lesion. Then urologists obtained sextant six-core SB. Each core was placed in an individual container and reported separately in accordance with the Ginsburg scheme. Histology was evaluated by senior uropathologists who were blinded to the imaging findings.
  Arms: 3TB+6SB group
Procedure: 3TB+12SB — The biopsy procedure was conducted by a highly skilled and experienced urologist who specializes in performing prostate biopsies. Prophylactic antibiotics were routinely used both before and one day prior to scheduled surgery. Each patient was placed in the left lateral position or lithotomy position. The ultrasound equipment used included a color Doppler ultrasound diagnostic instrument (Hitachi HiVision, Philips Epiq 7), transrectal probes, and corresponding puncture needle guns. Color Doppler examination was performed from the base to the apex. Urologists firstly obtained three-core TB from the lesion within the mpMRI suspicious lesion. Then urologists obtained fore-zone 12-core SB. Each core was placed in an individual container and reported separately in accordance with the Ginsburg scheme. Histology was evaluated by senior uropathologists who were blinded to the imaging findings.
  Arms: 3TB+12SB group

SUMMARY:
The goal of this randomized controlled trial (RCT) is to evaluate the efficacy and safety of different prostate biopsy schemes, including targeted biopsy plus sextant biopsy (3TB+6SB) and combination of targeted biopsy and 12-core systematic biopsy (3TB+12SB).

The main questions it aims to answer are:

Does 3TB+6SB promote the accurate diagnosis of clinically significant prostate cancer? What's the value of 3TB+6SB in improving the safety of prostate biopsy? Researchers will compare the cancer detection rates of 3TB+6SB and combination of 3TB+12SB to explore the efficacy of different prostate biopsy schemes. They will evaluate the safety profile of different prostate biopsy schemes through the complication rates and postoperative quality of life.

Participants will:

Receive 3TB+6SB or 3TB+12SB.

DETAILED DESCRIPTION:
Currently, combination of targeted biopsy and 12-core systematic biopsy (3TB+12SB) has been recommended for the diagnosis of patients with suspicious lesion found on multiparametric magnetic resonance imaging (mpMRI). Although the 3TB+12SB approach could effectively detect clinically significant prostate cancer (csPCa), the increased number of biopsy cores would increase the risk of complications and decrease the postoperative quality of life. In recent years, urological and radiologic thinking has changed after realizing that systemic biopsies may be reduced when the chance of missing a clinically significant lesion is low. More and more radiologists and urologists focused on the issue of optimization of prostate biopsy schemes. Some retrospective studies have proved that the cancer detection rate of targeted biopsy plus sextant biopsy (3TB+6SB) was not inferior to 3TB+12SB. However, the safety profile warrants further evaluation, and there is still a lack of high-quality, prospective evidence for the 3TB+6SB schemes. Thus, this randomized controlled trial (RCT) aims to evaluate the efficacy and safety of 3TB+6SB schemes and the routine 3TB+12SB schemes, provide high-quality evidence for the optimization of prostate biopsy schemes.

The main questions it aims to answer are:

Does 3TB+6SB promote the accurate diagnosis of clinically significant prostate cancer? What is the value of 3TB+6SB in improving the safety of prostate biopsy? This prospective RCT compared the csPCa detection rates of 3TB+6SB and 3TB+12SB. Participants were prospectively enrolled at Peking University First Hospital (Beijing, China) from September 2024 to February 2025. Participants were randomly allocated to 3TB+6SB group and 3TB+12SB group.

Researchers will compare the cancer detection rates of 3TB+6SB and 3TB+12SB to explore the efficacy of different prostate biopsy schemes. They will evaluate the safety profile of different prostate biopsy schemes through the complication rates and postoperative quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The age of the patient is between 45 and 85 years.
* No previous biopsy.
* Patients with single suspicious lesion, complete multiparametric magnetic resonance imaging (mpMRI) data, qualified image quality control, suspicious lesions, and Prostate Imaging Reporting and Data System version 2.1 (PI-RADS V2.1) of ≥ 3.
* Patients were in accordance with the indication of prostate biopsy, including patients with suspicious prostate nodes found by digital rectal examination (DRE), the suspicious lesions found by transrectal ultrasound (TRUS) or MRI, total prostate-specific antigen (tPSA) >10ng/mL, tPSA 4-10ng/mL with free-to-total PSA ratio (f/tPSA) <0.16 or PSA density (PSAD) >0.15.
* The prostate biopsy pathological results were complete. The time interval between prostate biopsy and prostate mpMRI examination should not exceed one month.
* Patients with complete clinical information.

Exclusion Criteria:

* The mpMRI data was unqualified or incomplete.
* Patients had received radiotherapy, chemotherapy, androgen deprivation therapy, or surgery treatment before prostate mpMRI examination or prostate biopsy.
* Patients with previous biopsy.
* Patients with PI-RADS V2.1 of < 3.
* Patients were not in accordance with the indication of prostate biopsy.
* The patient could not cooperate to complete the prostate biopsy.
* The patients or their family members refused to participate in this study.
* Patients with incomplete clinical information.

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The clinically significant prostate cancer (csPCa) detection rate | One month after the biopsy procedure.
  csPCa was defined as PCa with a grade group > 2 or GS ≥ 7. The reference standard was the pathological result.

SECONDARY OUTCOMES:
The overall complication rate | One week and one month after the biopsy procedure.
  The complication (mainly including bleeding, infection, pain, and lower urinary tract symptoms) rate after the prostate biopsy (3TB+6SB or 3TB+12SB).
The self-reported quality of life after the prostate biopsy | One week and one month after the biopsy procedure.
  The self-reported levels of pain and discomfort after the prostate biopsy was measured through visual analogue scale (VAS). The minimum and maximum values of VAS are 0 and 10. The higher VAS means the higher level of pain and discomfort.
The operation time of prostate biopsy | During the prostate biopsy procedure.
  The operation time of prostate biopsy was defined as the time from the beginning to the end of the prostate biopsy.
The PCa detection rate | One month after the biopsy procedure.
  The PCa detection rate for 3TB+6SB and 3TB+12SB.
The clinically insignificant PCa detection rate | One month after the biopsy procedure.
  The clinically insignificant PCa was defined as PCa with a grade group < 2 or GS < 7. The reference standard was the pathological result.
The Gleason score (GS) of the biopsy sample | One month after the biopsy procedure.
  The Gleason score (GS) was reported by senior uropathologists according to the Standards of Reporting for MRI Targeted Biopsy Studies (START) criteria and interpreted according to the recommendations of the International Society of Urological Pathology (ISUP) Grade Group. The minimum and maximum of GS are 3 and 5. The higher GS means the higher pathological grade.
The GS of radical prostatectomy (RP) specimens | One month after the biopsy procedure.
  For the RP specimens, the Gleason score (GS) was reported by senior uropathologists according to the Standards of Reporting for MRI Targeted Biopsy Studies (START) criteria and interpreted according to the recommendations of the International Society of Urological Pathology (ISUP) Grade Group. The minimum and maximum of GS are 3 and 5. The higher GS means the higher pathological grade.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Liu, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China